CLINICAL TRIAL: NCT05189964
Title: Total Hip Arthroplasty and Physical Activity in Patients Younger Than 50 Years
Acronym: THA&PA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: THA&PA
Record Dates: First submitted 2021-12-21; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Hip Osteoarthritis; Physical Inactivity
MeSH Terms: conditions — Osteoarthritis, Hip; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: THA is a widely applied procedure for osteoarthritis of the hip. After THA, one can expect an increase in physical activity due to the reduction of pain and increased range of motion of the hip joint, especially in young patients who in general have more active lifestyles. However, these young patients and their doctors don't know which increase in physical activity can be expected.

Objective: To measure the difference in physical activity before and after THA. Study design: Longitudinal prospective single center observational study. Study population: 87 patients who have primary THA under the age of 50 years. Excluding patients with an underlying oncologic disease which results in THA.

Intervention: N.a. Main study parameters/endpoints: The first primary endpoint is physical activity in minutes per day. The other primary endpoint is MVPA in minutes per day. Secondary endpoints are difference of TUG outcomes in seconds and the difference of 6MWT outcomes in meters. For the patients experience, the COPM total scores and NRS pain scores will be measured.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study requires three outpatient clinic visits. These visits will coincide with regular outpatient clinic visits, so patients will not have to come in extra for this study. During the preoperative and 1 year postoperative visit, the patients will complete the COPM. The patient will wear a PA monitor for 7 days after each visit. Patients might experience confronting feelings while being exposed to their PA activity profile after the study or experience mild discomfort while wearing the PA monitor since it will be worn 24 hours per day for 7 days. Also, filling in the questionnaires will take some time (5-10 minutes per questionnaire series). There are no significant physical risks associated to this study.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patient is between 16 and 50 years.
* The patient has an indication for primary THA.

Exclusion Criteria:

* Patients with an underlying oncologic disease which results in THA.
* Patients who are not able to walk.

Ages: 16 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients will be included from the patient population of the department of orthopaedics at the Radboudumc. Per year, approximately 80 patients under age of 50 years receive THA in this institute. The patient population has a male/female ratio of approximately 1:1.3, with multiple underlying diseases resulting in THA.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from time spent active in minutes per day | preoperative, 3 months postoperative, 12 months postoperative
Change from MVPA in minutes per day | preoperative, 3 months postoperative, 12 months postoperative

SECONDARY OUTCOMES:
TUG | preoperative, 3 months postoperative, 12 months postoperative
  Timed Up & Go
6MWT | preoperative, 3 months postoperative, 12 months postoperative
  6 minute walking test
COPM | preoperative, 12 months postoperative
  Canadian Occupational Performance Measure total scores

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided